CLINICAL TRIAL: NCT05581082
Title: Understanding Changes in Physical Function Using Principles of Precision Medicine
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 22-1230
Record Dates: First submitted 2022-09-21; First posted 2022-10-14 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Routine Clinical Care with PCP: All individuals will be seen by their primary care physician (PCP) in Geriatric Clinic. Patients previously diagnosed with frailty per their PCP. Their PCP visit will include independent assessment and physical therapy referral, and will begin a physical therapy-based strengthening intervention. Patients will be independently managed (assessment and intervention) by a Physical Therapist (PT). The PT will initiate an intervention plan (e.g., education and exercise)
  Interventions: Other: Pragmatic, exploratory study of Precision Medicine

INTERVENTIONS:
Other: Pragmatic, exploratory study of Precision Medicine — This pragmatic, exploratory study consists of individuals with frailty who are referred from routine care to a physical therapy-based strengthening intervention. This specific study will collect ancillary measures to evaluate our outcomes. The study staff will not be conducting any interventions themselves - the physical therapy program is as per usual care.

SUMMARY:
This is a pilot, feasibility study and the purpose of this study is exploratory. The goal is to provide the PI and study team with data using metabolomics that can be used to: a) demonstrate an ability to use such data in a future grant application; b) obtain data that determines the relationship between changes in physical function (objective and subjective) and potential metabolites.

DETAILED DESCRIPTION:
A pre/post, non-randomized, single-arm pilot natural clinical experiment trial of older adults (patients of UNC's Geriatrics Medicine Specialty Clinic, N=18) who will enroll in a physical therapy program as recommended by their primary care clinician. This pragmatic assessment consists of obtaining routine care data from the physical therapy visits and collecting blood to harness metabolomics data that can be used to: a) demonstrate an ability to use and analyze such data for a future grant application; b) determine the relationship between change in physical function and metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Older adults ≥65 years (of all genders and sexes) with diagnosis of frailty based on the Fried phenotype A UNC Geriatrics Medicine Specialty clinic at the Eastowne Clinic patient who has been referred for physical therapy to Elderfit;
* >2 Chronic medical conditions -these are based on the 21 Medicare multiple chronic conditions (e.g., alcohol abuse, Alzheimer's disease and related dementia, arthritis (osteoarthritis, rheumatoid), asthma, atrial fibrillation, autism spectrum disorders, cancer (breast, colorectal, lung, prostate), chronic kidney disease, chronic obstructive pulmonary disease, depression, diabetes, drug/substance abuse, heart failure, hepatitis, HIV/AIDS, hyperlipidemia, hypertension, ischemic heart disease, osteoporosis, schizophrenia/other psychotic disorders, stroke);
* Callahan cognitive screen ≥3 - this is a measure routinely used for clinical research in older adults. A screen of ≥3 suggests capacity to consent

Exclusion Criteria:

* Age <65 years;
* A medical diagnosis of dementia - all participants are required to have the ability to engage in the physical therapy-based intervention, complete questionnaires, and interact with others, all of which may be challenging in individuals with cognitive impairment;
* Individuals with life-threatening or untreated psychiatric diagnosis that would interfere with study participation and require significant modification to meet their needs such as untreated major depressive disorder, substance abuse, suicidal ideation or untreated severe mental illness (schizophrenia, bipolar disorder);
* Life-threatening illness including those receiving palliative care or hospice services;
* Individuals unwilling/unable to provide consent;
* Current participation in another physical therapy-based research study or program;
* Inability to complete the protocol procedures;
* Elective surgery in the next six months;
* Co-morbidities including: hospitalization for heart failure in past 6 months, history of advanced non-skin cancer (Stage III or IV); Advanced liver failure; Chronic renal insufficiency on hemodialysis;

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The investigators aim to screen 35 patients in the clinic (40% ineligible + 15% drop out) to complete 18 participants.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in blood sample | Up to 12 weeks
  The team will collect a blood sample at baseline (0- weeks) and follow-up (12-weeks) to conduct an untargeted metabolomic analysis to demonstrate potential peaks of protein within the blood reported in mg/dL.
Change in serum sample | Up to 12 weeks
  The team will collect a blood sample at baseline (0- weeks) and follow-up (12-weeks) to conduct an untargeted metabolomic analysis to demonstrate potential peaks of protein within the blood reported in g/dL.
Patient Reported Outcome Measure Information System-Global Health Questionnaire used to determine changes in Physical Function | Up to 12 weeks
  Providers will use the Patient Reported Outcome Measure Information System-Global Health Questionnaire to gauge physical, mental, and social aspects of health (5-point scale) to record the changes in physical function prior and after beginning the physical-therapy based program. A mean standardized score for the population is 50; 10 points indicate one standard deviation. Higher scores indicate better health.
Pittsburgh Fatigability Scale used to determine changes in Physical Function | Up to 12 weeks
  Providers will use the Pittsburgh Fatigability Scale will measure the fatigue of each sedentary, social, lifestyle, and physical activities to record the changes in physical function prior and after beginning the physical-therapy based program. 10 items total for physical and mental fatigue are summed to create two separate continuous scores, each ranging from 0 to 50. Higher scores indicate greater perceived physical or mental fatigability
Patient Activation Measure Survey used to determine changes in Physical Function | Up to 12 weeks
  Providers will use the Patient Activation Measure Survey will assess knowledge, skills, and confidence for managing health revealing insights into motivators, behaviors, attitudes, and outcomes to record the changes in physical function prior and after beginning the physical-therapy based program. An interval-level scale from 0-100. A lower patient activation score indicates a patient who is less active in managing their health, whereas a higher patient activation score indicates a patient who is more active in managing their health.
Saint Louis University Mental Status Examination Questionnaire used to determine changes in Physical Function | Up to 12 weeks
  Providers will use Saint Louis University Mental Status Examination to test orientation, memory, attention, and executive function, with items such as animal naming, digit span, figure recognition, clock drawing and size differentiation to record the changes in physical function prior and after beginning the physical-therapy based program (30-point, 11 questions total) Scores of 27 to 30 are considered normal in a person with a high school education. Scores between 21 and 26 suggest a mild neurocognitive disorder. Scores between 0 and 20 indicate dementia.
Community Healthy Activities Model Program for Senior Questionnaire used to determine changes in Physical Function | Up to 12 weeks
  Providers will use Community Healthy Activities Model Program for Senior Questionnaire to assesses weekly frequency and duration of various physical activities typically undertaken by older adults. Four different scores can be derived from the questionnaire: frequency of moderate or greater activity (MET >3.0, a composite score that ranges from 0 to 40, with higher scores indicating better performance); frequency of all physical activity (light, moderate, and vigorous); caloric expenditure of moderate or greater activity (light, moderate, vigorous); caloric expenditure of moderate or great activity; caloric expenditure of all physical activity.
Brief Resilience Scale used to determine changes in Physical Function | Up to 12 weeks
  Providers will use the Brief Resilience Scale to assess the ability to bounce back or recover from stress in order to record the changes in physical function prior and after beginning the physical-therapy based program. 6 total questions, scoring is on a range of 1-5. Once all six statements have been assessed, the total of the number is taken. This summing up will give an overall resilience score of between 6 and 30. Lower scores indicate lower levels of resilience.
Rapid Eating Assessment for Participants used to determine changes in Physical Function | Up to 12 weeks
  Providers will use Rapid Eating Assessment for Participants to perform a brief assessment of diet and physical activity to record the changes in physical function prior and after beginning the physical-therapy based program (Total scores range from 13 to 39 --higher quantities represent dietary quality characterized by optimal intake of fruits, vegetables, and whole grains and decreased intake of sugary foods, processed meats, and fried foods).
Patient Health Questionnaire used to determine changes in Physical Function | Up to 12 weeks
  Providers will use the Patient Health Questionnaire to identify signs or symptoms of depression to record the changes in physical function prior and after beginning the physical-therapy based program (9 questions total, ≤ 4 The score suggests the patient may not need depression treatment, >5-14 along with physician clinical judgment about treatment, based on patient's duration of symptoms and functional impairment, ≥ 15 Warrants treatment for depression, using antidepressant, psychotherapy and/or a combination of treatment).
Gait Speed used to determine changes in Physical Health. | Up to 12 weeks
  Providers will use gait speed to assess a comfortable gait speed for the patient to determine changes in physical health. Scale: healthy women aged 70-79 years is 1.13 meters per second (m/s) and for men 1.26 m/s. For women and men aged 80-99 the values are 0.94 meters per second (m/s) and 0.97 meters per second (m/s), respectively.
Grip Strength used to determine changes in Physical Health | Up to 12 weeks
  Providers will use grip strength to assess a comfortable gait speed for the patient to determine changes in physical health. Scale: Optimal cut-points were 24.9 kg for men 65-74 years, 20.8 kg for men 75-90 years, 15.2 kg for women 65-74 years, and 13.5 kg for women 75-90 years.

CONTACTS AND LOCATIONS:
Overall Officials: John Batsis, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States